CLINICAL TRIAL: NCT02422303
Title: Effects of Low Dose Ketamine Given at Induction of Anesthesia on Postoperative Mood in Patients With Depressive Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20150248H
Record Dates: First submitted 2015-04-16; First posted 2015-04-21 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2016-09

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Depression; Gynecoligical surgery; Ketamine
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine Group (Active Comparator): This group will receive ketamine 0.5mg/kg IV at induction of general anesthesia.
  Interventions: Drug: ketamine
- No ketamine group (No Intervention): This group will not receive ketamine at induction of general anesthesia.

INTERVENTIONS:
Drug: ketamine — Ketamine 0.5mg/kg will be given intravenously to group A at induction of general anesthesia.
  Other Names: ketalar
  Arms: Ketamine Group

SUMMARY:
Ketamine has been shown to have an antidepressant effect when given intravenously in doses of 2mg/kg. Ketamine is used as a standard induction drug during general anesthesia. It is known in this instance to decrease postoperative pain. No one has studied whether or not ketamine when given in doses used during general anesthesia (0.5mg/kg intravenous) has an antidepressant effect on surgical patients who suffer from depression. The study is designed to determine whether or not a small dose of ketamine when given at the induction of anesthesia could have an antidepressant effect on surgical patients with depression.

DETAILED DESCRIPTION:
Non-pregnant females between the ages of 18-65 who are being admitted for gynecological surgery will be given a bedside Goldberg depression screen as part of their routine preanesthetic assessment. If the patient scores five or above on the Goldberg depression screening, they will be asked if they would like to enroll in the study. Exclusion criteria include uncontrolled hypertension, pregnancy, or allergy to ketamine.

Once the patient is consented they will be randomized to one of two groups. Every patient will receive an antianxiety medication Midazolam and a narcotic fentanyl prior to going to the operating room. Group A will receive ketamine 0.5mg/kg intravenous as part of their induction for general anesthesia. Group B will not receive ketamine as part of their anesthetic. All other induction drugs will be at the discretion of the anesthesiologist performing the anesthetic.

The patients will be seen by a separate anesthesia provider (who is blinded to the group the patient is in) and the results of the depression screening will be added to the patient's data sheet.

The patients will be followed again one week after their surgery either in their hospital room (if still hospitalized) or by phone. They will again be given the Goldberg Depression screen and the data will again be added to their data sheet.

Several times during the study and at its conclusion the data will be matched with the patients group in order to assess for adverse events such as suicidal ideations, nausea and vomiting. If adverse events are noted, the study design will be altered to take into account the adverse events.

ELIGIBILITY:
Inclusion Criteria:

* History of or current depression scoring five or above on Goldberg Depression Screen

Exclusion Criteria:

* Uncontrolled hypertension, allergy to ketamine,pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonny C Gillis, M.D., Principal Investigator — Department of Anesthesiology UTHSCSA
Locations (1):
- University Hospital, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Naughton M, Clarke G, O'Leary OF, Cryan JF, Dinan TG. A review of ketamine in affective disorders: current evidence of clinical efficacy, limitations of use and pre-clinical evidence on proposed mechanisms of action. J Affect Disord. 2014 Mar;156:24-35. doi: 10.1016/j.jad.2013.11.014. Epub 2013 Dec 10. PMID 24388038
- [Background] Martinowich K, Jimenez DV, Zarate CA Jr, Manji HK. Rapid antidepressant effects: moving right along. Mol Psychiatry. 2013 Aug;18(8):856-63. doi: 10.1038/mp.2013.55. Epub 2013 May 21. PMID 23689537

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ketamine Group | No Ketamine Group
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Group | No Ketamine Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Depression Score Using Goldberg Depression Screening Test
Description: The Goldberg screening test consists of 18 questions which are answered based upon the previous 10-14 days to assess depression:
  0-not at all
  1. just a little
  2. somewhat
  3. moderately
  4. quite a lot
  5. very much
  The scores are summed, and the ranges are assessed:
  0 - 9 No depression likely 10 - 21 Possible symptoms that may be due to depression or other medical issues.
  22 - 35 Mild to Moderate Depression. 36 - 53 Moderate to Severe Depression 54 and up Severely Depressed The higher the score, the more severe you depression is likely to be.
Time Frame: One week
Population: Participant data were destroyed at study termination, and no analysis was performed, since no longer available.
Arm/Group | Ketamine Group | No Ketamine Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ketamine Group | No Ketamine Group
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes